CLINICAL TRIAL: NCT00260208
Title: A Multicenter, Randomized, Open-label Study to Compare the Development of Liver Fibrosis at 12 Months After Transplantation for Hepatitis C Cirrhosis in Patients Receiving Either Cyclosporine Microemulsion or Tacrolimus
Brief Title: Liver Fibrosis in Patients Transplanted for Hepatitis C Receiving Either Cyclosporine Microemulsion or Tacrolimus
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was prematurely terminated due to poor recruitment.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COLO400A2426
Record Dates: First submitted 2005-11-30; First posted 2005-12-01 (Estimated); Results first posted 2011-10-26 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Liver Transplant; Hepatitis C
Keywords: Liver transplant, adults, hepatitis C, liver fibrosis, cyclosporine microemulsion, tacrolimus
MeSH Terms: conditions — Hepatitis C; Liver Cirrhosis | interventions — Cyclosporine; Tacrolimus

ARMS (2):
- Cyclosporin A (Active Comparator): The first administration of Cyclosporin A (CsA) was within the first 24 hours post-transplantation at an initial dose of 10-15mg/kg/day either orally, via a nasogastric (NG) tube or intravenously (i.v). Twice daily (b.i.d.) administration was maintained throughout the study period. During the study, the dose of CsA was adjusted, as necessary, to achieve and maintain the C2 or C0 blood CsA concentration within the target ranges.
  Before enrolling the first patient, each center chose the adjunct immunosuppressive (IS) regimen between:
  * Steroids administered and tapered as per local practice
  * interleukin-2 receptor (IL-2R) antagonists + mycophenolic acid (MPA): Induction with IL-2R antagonists; Dosages were as per center practice. Patients received mycophenolic acid (MPA) no later than 24 hours after reperfusion of the graft. Dosages were as per local practice.
  The regimen selected by the center was to be given to all patients enrolled in the trial from this center.
  Interventions: Drug: Cyclosporine A
- Tacrolimus (Active Comparator): Tacrolimus was administered within the first 24 hours post-transplantation at an initial dose of 0.1-0.15 mg/kg/day in 2 divided doses (twice daily at 12-hour interval) either orally or via a nasogastric (NG) tube or intravenously (i.v). Twice daily (b.i.d.) administration was maintained throughout study period. Throughout the study, the dose of tacrolimus was adjusted as necessary to achieve and maintain C0 tacrolimus concentrations within target ranges.
  Before enrolling the first patient, each center chose adjunct immunosuppressive (IS) regimen between:
  * Steroids administered and tapered as per local practice
  * interleukin-2 receptor (IL-2R) antagonists + mycophenolic acid (MPA): Induction with IL-2R antagonists; Dosages were as per center practice. Patients received mycophenolic acid (MPA) no later than 24 hours after reperfusion of the graft. Dosages were as per local practice.
  The regimen selected by center was to be given to all patients enrolled in trial from this center.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Cyclosporine A — Initial dose of 10-15mg/kg/day either orally, via a nasogastric (NG) tube or intravenously (i.v.) within the first 24 hours post-transplantation.
  Other Names: Neoral
  Arms: Cyclosporin A
Drug: Tacrolimus — Tacrolimus was administered within the first 24 hours post-transplantation at an initial dose of 0.1-0.15 mg/kg/day in 2 divided doses either orally or via a nasogastric (NG) tube or intravenously (i.v).
  Arms: Tacrolimus

SUMMARY:
Following a transplant for hepatitis C cirrhosis, the infection comes back in 70-90% of cases and over time causes fibrosis and eventually cirrhosis of the new liver. The aim of this study was to see if the frequency of liver fibrosis was different with cyclosporine microemulsion than tacrolimus

ELIGIBILITY:
Inclusion criteria

* Reason for transplant is end-stage liver disease due to hepatitis C cirrhosis
* Patients receiving a first liver transplant from a deceased or living donor
* Patients in whom biopsies will be possible

Exclusion criteria

* Recipients of a liver from an hepatitis C virus positive (HCV+), human immunodeficiency virus positive (HIV+) or hepatitis B virus positive (HBV+) donor
* Patients with any severe coexisting disease or suffering any unstable medical condition or co-infected with HBV or HIV
* Patients with co-existing alcoholic disease who have not been abstinent for at least 6 months
* Transplanted for liver cancer exceeding a pre-defined size
* Pregnant or nursing women

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2006-01; Primary Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Investigative Site, East Hanover, New Jersey, United States
- Novartis Investigational Site, Zurich, Switzerland

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 361 patients were randomized, 185 to the cyclosporin A arm and 176 to tacrolimus. Five patients (1 cyclosporine A, 4 tacrolimus) did not receive any dose of study medication and were therefore excluded from the safety population.
Groups:
- Cyclosporin A: The first administration of Cyclosporin A (CsA) was within the first 24 hours post-transplantation at an initial dose of 10-15mg/kg/day in 2 divided doses (twice daily at 12-hour interval) either orally, via a nasogastric (NG) tube or intravenously (i.v). Twice daily (b.i.d.) administration was maintained throughout the study period. During the study, it was recommended that the dose of CsA was adjusted, as necessary, to achieve and maintain the C2 or C0 blood CsA concentration within the target ranges.
- Tacrolimus: Tacrolimus was administered within the first 24 hours post-transplantation at an initial dose of 0.1-0.15 mg/kg/day in 2 divided doses (twice daily at 12-hour interval) either orally or via a nasogastric (NG) tube or intravenously (i.v). Twice daily (b.i.d.) administration was maintained throughout the study period. During the course of the study, the dose of tacrolimus was adjusted as necessary to achieve and maintain the C0 tacrolimus concentrations within target ranges.
Period: Overall Study
Arm/Group | Cyclosporin A | Tacrolimus
Started | 184 ("Started" indicates safety population.) | 172
Intent to Treat (ITT) Population | 182 | 169
Modified ITT | 101 | 96
Completed | 137 | 138
Not Completed | 47 | 34
Not completed — Subject withdrew consent | 11 | 7
Not completed — Lost to Follow-up | 6 | 1
Not completed — Death | 12 | 10
Not completed — Missing | 18 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cyclosporin A | Tacrolimus | Total
Number analyzed (Participants) | 182 | 169 | 351
Age Continuous [Mean (Standard Deviation); unit: years] — Baseline measurements were based on intent-to-treat population which included all patients as randomized that were transplanted, received at least one dose of study drug and had at least one post-baseline efficacy assessment.
  years | 54.4 (6.9) | 54.4 (7.1) | 54.4 (7.0)
Age, Customized [Number; unit: Participants]
  < 65 years | 163 | 154 | 317
  ≥ 65 years | 19 | 15 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 48 | 105
  Male | 125 | 121 | 246

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Fibrosis Score 2 or Above [Ishak-Knodell Fibrosis Score (FS) ≥ 2] Within 1 Year Post-transplant
Description: Assessment of hepatic fibrosis was performed with liver biopsies at Day 1, Month 6, 12 and 24, read centrally by two independent pathologists blinded to treatment arm and time of biopsy. Ishak-Knodell score was used to stage liver disease; 0= None; 1= Portal fibrosis (some); 2= Portal fibrosis (most); 3= Bridging fibrosis (few); 4= Bridging fibrosis (many); 5 = Incomplete cirrhosis; 6 = Cirrhosis. Higher score indicates greater fibrosis. Logistic regression on the presence of IK>=2 was applied based on central biopsy readings only.
Time Frame: 1 year post-transplant
Population: The modified intent-to-treat population (mITT) included patients treated with study drug at least up to 30 days before Month 12 visit and a liver biopsy had to be performed at this visit. Also included were patients with an earlier biopsy that showed an Ishak-Knodell fibrosis score ≥2 and treated at least up to 30 days before that biopsy was taken.
Measure: Number; unit: Participants
Arm/Group | Cyclosporin A | Tacrolimus
Number analyzed (Participants) | 88 | 77
Participants | 63 | 52

2. Secondary Outcome: Number of Participants With Combined Endpoint of Death or Graft Loss or Fibrosis Score (FS) ≥ 2
Description: The number of participants with combined end point of death or graft loss or presented with a Ishak-Knodell fibrosis score (FS) ≥2 was calculated. Graft loss was considered to have occurred when allograft was presumed to be lost if a patient had liver retransplant or died. Assessment of hepatic fibrosis was performed with liver biopsies read centrally. Ishak-Knodell FS was used to stage liver disease; 0=none; 1=portal fibrosis (some); 2=portal fibrosis (most); 3=bridging fibrosis (few); 4=bridging fibrosis (many); 5=Incomplete cirrhosis; 6=cirrhosis. Higher score indicates greater fibrosis.
Time Frame: 1 year post-transplant
Population: Intent-to-treat (ITT) population: all patients as randomized that were transplanted, received at least one dose of study drug and had at least one post-baseline efficacy assessment.
Measure: Number; unit: Participants
Arm/Group | Cyclosporin A | Tacrolimus
Number analyzed (Participants) | 182 | 169
Participants | 77 | 71

3. Secondary Outcome: Number of Participants With Fibrosing Cholestatic Hepatitis
Description: Fibrosing cholestatic hepatitis (FCH) is characterized by progressive jaundice with a rapid decline in liver function leading to liver failure, most often associated with markedly elevated viral levels detected in the bloodstream (e.g. more than 20 times pre-liver transplantation levels) and in the liver tissue as well. The presence of FCH was reported based on the diagnosis given by the investigator.
Time Frame: 1 year post-transplantation
Population: Intent-to-treat population: all patients as randomized that were transplanted, received at least one dose of study drug and had at least one post-baseline efficacy assessment.
Measure: Number; unit: Participants
Arm/Group | Cyclosporin A | Tacrolimus
Number analyzed (Participants) | 182 | 169
Participants | 9 | 6

4. Secondary Outcome: Number of Participants With Death, Graft Loss, Death or Graft Loss, Graft Loss With Re-transplantation
Description: Graft loss was considered to have occurred when allograft was presumed to be lost if a patient had a liver re-transplant or died.
Time Frame: 1 year post-transplant
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Cyclosporin A | Tacrolimus
Number analyzed (Participants) | 182 | 169
Participants
  Death | 15 | 15
  Graft loss | 8 | 13
  Death or Graft loss | 19 | 23
  Graft loss with re-transplantation | 3 | 8

5. Secondary Outcome: Number of Participants With Treated Acute Rejection, Biopsy Proven Acute Rejection (BPAR), and Sub-clinical Rejection
Description: Treated acute rejection is defined as an acute rejection, clinically suspected, whether biopsy-proven or not, which has been treated and confirmed by the investigator according to the response to therapy. BPAR was defined as a treated acute rejection confirmed by biopsy. The local pathologist graded biopsies according to the Banff (1997) criteria. A sub-clinical rejection was defined as a rejection identified by center driven biopsy, i.e. a biopsy performed routinely at some pre-defined time points after transplantation as per center practice in the absence of any clinical signs of rejection.
Time Frame: 1 year post-transplant
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Cyclosporin A | Tacrolimus
Number analyzed (Participants) | 182 | 169
Participants
  Treated acute rejection | 28 | 22
  Biopsy prove acute rejection (BPAR) | 28 | 19
  Sub-clinical rejection | 4 | 4

6. Secondary Outcome: Number of Participants With Combined Endpoint of Death or Graft Loss or Biopsy Proven Acute Rejection (BPAR)
Description: BPAR was defined as a treated acute rejection confirmed by biopsy. The local pathologist graded biopsies according to the Banff (1997) criteria. Graft loss was considered to have occurred when allograft was presumed to be lost if a patient had a liver re-transplant or died.
Time Frame: 1 year post-transplant
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Cyclosporin A | Tacrolimus
Number analyzed (Participants) | 182 | 169
Participants | 45 | 42

7. Secondary Outcome: Number of Participants With Death or Re-transplantation Due to Recurrence of Hepatitis C Cirrhosis
Description: Cirrhosis was resulted due to the recurrence of the hepatitis C virus infection in the transplanted liver.
Time Frame: 1 year post-transplant
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Cyclosporin A | Tacrolimus
Number analyzed (Participants) | 182 | 169
Participants | 16 | 17

8. Secondary Outcome: Number of Participants With Fibrosis Score 2 or Above [Ishak-Knodell Fibrosis Score (FS) ≥ 2] Within 1 Year Post-transplant (Intent to Treat Population)
Description: Assessment of hepatic fibrosis was performed with liver biopsies at Day 1, Month 6, 12 and 24, read centrally by two independent pathologists blinded to treatment arm and time of biopsy. Ishak-Knodell score was used to stage liver disease; 0= None; 1= Portal fibrosis (some); 2= Portal fibrosis (most); 3= Bridging fibrosis (few); 4= Bridging fibrosis (many); 5 = Incomplete cirrhosis; 6 = Cirrhosis. Higher score indicates greater fibrosis.
Time Frame: 1 year post-transplant
Population: The Intent-To-Treat (ITT) population consisted of all patients as randomized that were transplanted, received at least one dose of study drug and had at least one post-baseline efficacy assessment.
Measure: Number; unit: Participants
Arm/Group | Cyclosporin A | Tacrolimus
Number analyzed (Participants) | 182 | 169
Participants | 63 | 54

9. Secondary Outcome: Mean Value of Liver Function Tests at 1 Year Post-transplantation
Description: The mean value (in Units per liter, IU/L) of following tests were calculated at 1 year post-transplant:
  * Serum glutamic pyruvic transaminase (SGPT)
  * Serum Glutamic Oxaloacetic Transaminase (SGOT)
  * Bilirubin
  * Alkaline Phosphate
  * γ-Glutamyltransferase (GGT)
Time Frame: 1 year post-transplant
Population: Intent-to-treat (ITT) population: all patients as randomized that were transplanted, received at least one dose of study drug and had at least one post-baseline efficacy assessment. "n" is number participants with assessable data in each category.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Cyclosporin A | Tacrolimus
Number analyzed (Participants) | 112 | 115
IU/L
  SGPT (n= 112, 112) | 100.5 (178.8) | 81.7 (82.5)
  SGOT (n= 112,112) | 92.0 (122.3) | 72.8 (98.2)
  Bilirubin (n= 111, 115) | 40.3 (85.5) | 19.3 (27.9)
  Alkaline Phosphate (n= 111, 115) | 174.7 (152.9) | 152.9 (127.3)
  GGT (n= 103, 110) | 182.2 (224.3) | 168.5 (278.7)

10. Secondary Outcome: Log-transformed Hepatitis C Virus Ribonucleic Acid (HCV RNA) Values up to 1 Year Post Transplant
Description: HCV RNA was measured (IU/µL)centrally pre-transplant (Day 1) and at 48 hours (Day 3), Day 8 and 29, Month 6 and 12 post-transplant and concomitantly to any additional biopsies performed.
Time Frame: Pre-transplant (Day 1), Day , Day 8, Day 29, Month 6 and 12 post- transplant
Population: Intent-to-treat (ITT) population: all patients as randomized that were transplanted, received at least one dose of study drug and had at least one post-baseline efficacy assessment. "n" in each of the categories is the number of participants with data at the given time point.
Measure: Mean (Standard Deviation); unit: IU/µL
Arm/Group | Cyclosporin A | Tacrolimus
Number analyzed (Participants) | 182 | 169
IU/µL
  Day 1 (n=116, 111) | 0.71 (0.887) | 0.62 (0.809)
  Day 3 (n= 136, 120) | 0.98 (1.112) | 0.91 (1.024)
  Day 8 (n= 122, 117) | 1.58 (1.569) | 1.45 (1.557)
  Day 29 (n=128, 109) | 2.56 (1.658) | 2.74 (1.439)
  Month 6 (n=96, 98) | 3.45 (1.069) | 3.14 (1.332)
  Month 12 (n= 85, 88) | 3.17 (1.246) | 3.13 (1.385)

11. Secondary Outcome: Percentage of Participants With an Increase of at Least 1 Stage in Fibrosis
Description: Assessment of hepatic fibrosis was performed with liver biopsies at Day 1, Month 6, 12 and 24, read centrally by two independent pathologists blinded to treatment arm and time of biopsy. Ishak-Knodell score was used to stage liver disease; 0= None; 1= Portal fibrosis (some); 2= Portal fibrosis (most); 3= Bridging fibrosis (few); 4= Bridging fibrosis (many); 5 = Incomplete cirrhosis; 6 = Cirrhosis. Higher score indicates greater fibrosis. An increase of at least 1 stage demonstrated a worsening of the disease, i.e. the transition from one score to the next higher one.
Time Frame: Between 1 and 2 years
Population: The outcome measure was not analyzed because of premature termination of study.
Measure: Number; unit: Percentage of participants
Arm/Group | Cyclosporin A | Tacrolimus
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Mean Fibrosis Score
Description: Assessment of hepatic fibrosis was performed with liver biopsies at Day 1, Month 6, 12 and 24, read centrally by two independent pathologists blinded to treatment arm and time of biopsy. Ishak-Knodell score was used to stage liver disease; 0= None; 1= Portal fibrosis (some); 2= Portal fibrosis (most); 3= Bridging fibrosis (few); 4= Bridging fibrosis (many); 5 = Incomplete cirrhosis; 6 = Cirrhosis. Higher score indicates greater fibrosis. The mean score was equivalent to mean of IK at 1 and 2 years (evolution over time).
Time Frame: At 1and 2 years and its evolution over time
Population: This outcome was not analyzed because of premature termination of study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cyclosporin A | Tacrolimus
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Cyclosporin A | Tacrolimus
Serious Adverse Events (participants affected / at risk) | 148/184 | 138/172
Other Adverse Events (participants affected / at risk) | 182/184 | 167/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclosporin A (N=184) | Tacrolimus (N=172)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 2
Cardiac disorder (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Abdominal adhesions (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 9
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2
Abdominal rigidity (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 2 | 2
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Duodenitis (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0
Faeces pale (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 1 | 2
Inguinal hernia (Gastrointestinal disorders) | 1 | 2
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Intestinal strangulation (Gastrointestinal disorders) | 1 | 0
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 0 | 4
Mechanical ileus (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 6 | 2
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Effusion (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 2
Hernia (General disorders) | 1 | 0
Hernia obstructive (General disorders) | 1 | 1
Hernia pain (General disorders) | 0 | 1
Impaired healing (General disorders) | 2 | 0
Multi-organ failure (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 13 | 9
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1
Bile duct necrosis (Hepatobiliary disorders) | 1 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 3
Bile duct stenosis (Hepatobiliary disorders) | 8 | 3
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Biliary cirrhosis (Hepatobiliary disorders) | 1 | 0
Biliary ischaemia (Hepatobiliary disorders) | 0 | 1
Biloma (Hepatobiliary disorders) | 1 | 2
Cholangitis (Hepatobiliary disorders) | 9 | 2
Cholestasis (Hepatobiliary disorders) | 1 | 1
Haemobilia (Hepatobiliary disorders) | 0 | 1
Hepatic artery stenosis (Hepatobiliary disorders) | 2 | 2
Hepatic artery thrombosis (Hepatobiliary disorders) | 1 | 3
Hepatic failure (Hepatobiliary disorders) | 5 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 3
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 1
Hepatic infiltration eosinophilic (Hepatobiliary disorders) | 0 | 1
Hepatic vein thrombosis (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatitis cholestatic (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Liver transplant rejection (Immune system disorders) | 11 | 7
Transplant rejection (Immune system disorders) | 2 | 2
Abdominal abscess (Infections and infestations) | 1 | 2
Abdominal sepsis (Infections and infestations) | 0 | 1
Abdominal wall abscess (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bone abscess (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Cytomegalovirus hepatitis (Infections and infestations) | 0 | 2
Cytomegalovirus infection (Infections and infestations) | 7 | 1
Cytomegalovirus viraemia (Infections and infestations) | 1 | 0
Enterobacter infection (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1
Groin abscess (Infections and infestations) | 1 | 0
Hepatic infection (Infections and infestations) | 1 | 0
Hepatitis C (Infections and infestations) | 77 | 65
Herpes zoster (Infections and infestations) | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Intervertebral discitis (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 3 | 0
Lung infection (Infections and infestations) | 0 | 1
Neurological infection (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Pericarditis fungal (Infections and infestations) | 0 | 1
Peritonitis bacterial (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 2 | 7
Pneumonia bacterial (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 8 | 5
Septic shock (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Tuberculosis liver (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 3
Wound infection (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Biliary anastomosis complication (Injury, poisoning and procedural complications) | 1 | 4
Chemical peritonitis (Injury, poisoning and procedural complications) | 2 | 0
Collapse of lung (Injury, poisoning and procedural complications) | 1 | 0
Complications of transplanted liver (Injury, poisoning and procedural complications) | 3 | 10
Gastrointestinal injury (Injury, poisoning and procedural complications) | 0 | 1
Graft loss (Injury, poisoning and procedural complications) | 1 | 1
Hepatic haematoma (Injury, poisoning and procedural complications) | 3 | 0
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 3 | 1
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1
Post procedural bile leak (Injury, poisoning and procedural complications) | 5 | 4
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 1
Postoperative fever (Injury, poisoning and procedural complications) | 1 | 0
Procedural site reaction (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 | 2
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Wound decomposition (Injury, poisoning and procedural complications) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 2
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 3 | 0
Blood pressure increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 2
Hepatitis C virus test positive (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 14 | 9
Transaminases increased (Investigations) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 4
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 2 | 1
Dizziness (Nervous system disorders) | 0 | 2
Encephalopathy (Nervous system disorders) | 2 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 1 | 1
Hypertensive encephalopathy (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1
Neurological symptom (Nervous system disorders) | 1 | 0
Neurotoxicity (Nervous system disorders) | 1 | 2
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Alcoholism (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 3 | 1
Psychotic disorder (Psychiatric disorders) | 2 | 0
Substance abuse (Psychiatric disorders) | 0 | 1
Transient psychosis (Psychiatric disorders) | 3 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 1
Anuria (Renal and urinary disorders) | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 6 | 3
Renal failure acute (Renal and urinary disorders) | 14 | 6
Renal impairment (Renal and urinary disorders) | 2 | 2
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Brain hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2
Haemodynamic instability (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 2 | 0
Intra-abdominal haematoma (Vascular disorders) | 1 | 0
Intra-abdominal haemorrhage (Vascular disorders) | 2 | 2
Malignant hypertension (Vascular disorders) | 1 | 1
Thrombosis (Vascular disorders) | 0 | 1
Venoocclusive disease (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclosporin A (N=184) | Tacrolimus (N=172)
Anaemia (Blood and lymphatic system disorders) | 51 | 54
Coagulopathy (Blood and lymphatic system disorders) | 3 | 9
Leukopenia (Blood and lymphatic system disorders) | 17 | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 23 | 28
Abdominal distension (Gastrointestinal disorders) | 14 | 7
Abdominal pain (Gastrointestinal disorders) | 31 | 44
Abdominal pain upper (Gastrointestinal disorders) | 9 | 14
Ascites (Gastrointestinal disorders) | 31 | 29
Constipation (Gastrointestinal disorders) | 64 | 62
Diarrhoea (Gastrointestinal disorders) | 41 | 57
Dyspepsia (Gastrointestinal disorders) | 15 | 14
Nausea (Gastrointestinal disorders) | 55 | 59
Vomiting (Gastrointestinal disorders) | 30 | 25
Asthenia (General disorders) | 15 | 9
Fatigue (General disorders) | 24 | 19
Generalised oedema (General disorders) | 12 | 12
Non-cardiac chest pain (General disorders) | 7 | 13
Oedema peripheral (General disorders) | 61 | 58
Pyrexia (General disorders) | 52 | 47
Bile duct stenosis (Hepatobiliary disorders) | 11 | 12
Cholestasis (Hepatobiliary disorders) | 10 | 10
Hyperbilirubinaemia (Hepatobiliary disorders) | 13 | 7
Cytomegalovirus infection (Infections and infestations) | 16 | 5
Hepatitis C (Infections and infestations) | 19 | 21
Nasopharyngitis (Infections and infestations) | 10 | 13
Pneumonia (Infections and infestations) | 6 | 15
Urinary tract infection (Infections and infestations) | 24 | 16
Incision site pain (Injury, poisoning and procedural complications) | 33 | 27
Post procedural bile leak (Injury, poisoning and procedural complications) | 8 | 9
Post procedural discharge (Injury, poisoning and procedural complications) | 6 | 10
Procedural pain (Injury, poisoning and procedural complications) | 50 | 59
Blood bilirubin increased (Investigations) | 15 | 6
Blood creatinine increased (Investigations) | 35 | 23
Blood glucose increased (Investigations) | 4 | 9
Blood potassium decreased (Investigations) | 10 | 9
Haemoglobin decreased (Investigations) | 8 | 11
Liver function test abnormal (Investigations) | 31 | 25
Urine output decreased (Investigations) | 17 | 16
Decreased appetite (Metabolism and nutrition disorders) | 21 | 16
Diabetes mellitus (Metabolism and nutrition disorders) | 26 | 28
Fluid overload (Metabolism and nutrition disorders) | 11 | 13
Hyperglycaemia (Metabolism and nutrition disorders) | 46 | 49
Hyperkalaemia (Metabolism and nutrition disorders) | 27 | 28
Hypoalbuminaemia (Metabolism and nutrition disorders) | 13 | 14
Hypocalcaemia (Metabolism and nutrition disorders) | 17 | 17
Hypokalaemia (Metabolism and nutrition disorders) | 33 | 29
Hypomagnesaemia (Metabolism and nutrition disorders) | 39 | 43
Hyponatraemia (Metabolism and nutrition disorders) | 11 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 38 | 25
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11 | 16
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 13 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 14
Dizziness (Nervous system disorders) | 8 | 11
Headache (Nervous system disorders) | 45 | 39
Tremor (Nervous system disorders) | 26 | 30
Agitation (Psychiatric disorders) | 16 | 24
Anxiety (Psychiatric disorders) | 30 | 21
Confusional state (Psychiatric disorders) | 9 | 15
Depression (Psychiatric disorders) | 17 | 16
Insomnia (Psychiatric disorders) | 65 | 64
Oliguria (Renal and urinary disorders) | 22 | 20
Renal failure (Renal and urinary disorders) | 19 | 18
Renal failure acute (Renal and urinary disorders) | 23 | 16
Renal impairment (Renal and urinary disorders) | 21 | 15
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 11 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 24
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 25 | 31
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 7 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 21 | 19
Rash (Skin and subcutaneous tissue disorders) | 11 | 5
Hypertension (Vascular disorders) | 92 | 69
Hypotension (Vascular disorders) | 20 | 15

LIMITATIONS AND CAVEATS:
This study was prematurely discontinued due to poor recruitment. Since only a small patient group could be analyzed for primary outcome measure, robust conclusions on the effect of the two calcineurin inhibitors on the fibrosis score cannot be drawn.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.